CLINICAL TRIAL: NCT03575403
Title: A Novel Drug Combination for Alcohol-Use Disorders: A Human Laboratory Study
Brief Title: Behavioral Effects of Drugs: Inpatient (36) (Alcohol, Duloxetine, and Methylphenidate)
Acronym: BED[IN]:36
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Craig Rush (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor-Investigator, Craig Rush, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Basic Science
Other Study IDs: 44796; R01AA026255 (NIH)
Record Dates: First submitted 2018-06-22; First posted 2018-07-02 (Actual); Results first posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2024-04

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Ethanol; Duloxetine Hydrochloride; Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Subjects received oral placebo capsules one time daily.
  Interventions: Drug: Alcohol; Drug: Placebos; Drug: Methylphenidate
- Duloxetine (60 MG) (Experimental): Subjects received 60 mg of oral duloxetine one time daily.
  Interventions: Drug: Duloxetine (60 MG)
- Duloxetine (30 MG) (Experimental): Subjects received 30 mg of oral duloxetine one time daily. Note: only 2 subjects were enrolled in this arm prior to the arm being removed in the summer of 2020. Data from this arm will not be reported in order to avoid any HIPAA violation due to the small number of subjects in this arm.
  Interventions: Drug: Duloxetine (30 MG)

INTERVENTIONS:
Drug: Alcohol — In each arm and during sessions, subjects will receive doses of alcohol designed to raise breath alcohol levels (BAL) to 0.03 g/dl.
  Arms: Placebo
Drug: Placebos — Subjects will receive oral placebo capsules.
  Arms: Placebo
Drug: Duloxetine (60 MG) — Subjects will receive 60-mg of oral duloxetine capsules.
  Arms: Duloxetine (60 MG)
Drug: Methylphenidate — Subjects will receive methylphenidate capsules.
  Arms: Placebo
Drug: Duloxetine (30 MG) — Subjects will receive 30-mg of oral duloxetine capsules.
  Arms: Duloxetine (30 MG)

SUMMARY:
This study will evaluate the behavioral effects of alcohol during maintenance on placebo, duloxetine, methylphenidate and duloxetine combined with methylphenidate using sophisticated human laboratory methods.

DETAILED DESCRIPTION:
Prior to the outbreak of the COVID-19 virus and subsequent work-from-home orders from the state of Kentucky government, participants completed five overnight sessions at theUniversity of Kentucky Inpatient Research Unit in the medical center. The protocol was then changed to have five sessions scheduled to be completed on an outpatient basis in the late afternoon/early evening. This protocol change was enacted following the resumption of research in the fall of 2020.

For both the inpatient and outpatient portions of this protocol, the first of these sessions was a practice session to familiarize participants with experimental procedures. The subsequent four experimental sessions were conducted following one-week maintenance on a methylphenidate dose (0, 20, 40, and 60 mg/day; within-subjects factor) over the span of four weeks. Participants were assigned to either an active duloxetine arm (60 mg/day) or placebo arm (between-subjects factor) also for the span of four weeks. The outcome measures collected were the same for both the inpatient and outpatient aspects of the study.

Subjects received 30 mg of oral duloxetine one time daily. Note: only 2 subjects were enrolled in this arm prior to the arm being removed in the summer of 2020. Data from this arm will not be reported in order to avoid any HIPAA violation due to the small number of subjects in this arm.

Please note that at the initial execution of the study, there were three duloxetine arms: 0, 30, and 60 mg/day. Two participants received 30 mg/day. However, visual inspection of their data revealed that their data was not appreciably different from participants in the 60 mg/day duloxetine arm. Therefore, we have added the data from these two participants to the 60 mg/day duloxetine arm for all reported data.

ELIGIBILITY:
Inclusion Criteria:

* able to speak/read English
* not seeking treatment at the time of the study
* one binge drinking episode (5+/4+ standard alcoholic drinks per drinking session for men and women, respectively) in the past 30 days
* recent alcohol use verified by ethyl glucuronide positive urine, as well as fulfillment of DSM-5 diagnostic criteria for alcohol use disorder
* ECG within normal limits
* otherwise healthy
* body mass index of 19-35
* females using an effective form of birth control and not pregnant or breast feeding
* judged by the medical staff to be psychiatrically and physically healthy
* able to abstain from alcohol for 12 hours prior to session

Exclusion Criteria

* Not under 21 years of age or over 55 years of age
* no contraindications/allergies to alcohol, duloxetine, or methylphenidate

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Rush, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Please note that at the initial execution of the study, there were three duloxetine arms: 0, 30, and 60 mg/day. Two participants received 30 mg/day. However, to avoid the risk of HIPAA violation, data from these two participants will not be reported.
Groups:
- Placebo: Subjects received oral placebo capsules one time daily.
  Alcohol: In each arm and during sessions, subjects will receive doses of alcohol designed to raise breath alcohol levels (BAL) to 0.03 g/dl.
  Placebos: Subjects will receive placebo capsules.
  Methylphenidate: Subjects will receive methylphenidate capsules.
- Duloxetine (30 MG): Subjects received 30 mg of oral duloxetine one time daily.
  Alcohol: In each arm and during sessions, subjects will receive doses of alcohol designed to raise breath alcohol levels (BAL) to 0.03 g/dl.
  Duloxetine: Subjects will receive duloxetine capsules.
  Methylphenidate: Subjects will receive methylphenidate capsules.
- Duloxetine (60 MG): Subjects received 60 mg of oral duloxetine one time daily.
  Alcohol: In each arm and during sessions, subjects will receive doses of alcohol designed to raise breath alcohol levels (BAL) to 0.03 g/dl.
  Duloxetine: Subjects will receive duloxetine capsules.
  Methylphenidate: Subjects will receive methylphenidate capsules.
Period: Overall Study
Arm/Group | Placebo | Duloxetine (30 MG) | Duloxetine (60 MG)
Started | 11 | 2 | 6
0 mg Methylphenidate | 11 | 2 | 6
20 mg Methylphenidate | 10 | 2 | 6
40 mg Methylphenidate | 10 | 2 | 6
60 mg Methylphenidate | 9 | 2 | 6
Completed | 9 | 2 | 6
Not Completed | 2 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — One subject left due to personal reasons unrelated to study-procedures | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Duloxetine (30 MG): Subjects received 30 mg of oral duloxetine one time daily.
  Alcohol: In each arm and during sessions, subjects will receive doses of alcohol designed to raise breath alcohol levels (BAL) to 0.03 g/dl.
  Duloxetine: Subjects will receive duloxetine capsules.
- Total: Total of all reporting groups
Arm/Group | Placebo | Duloxetine (30 MG) | Duloxetine (60 MG) | Total
Number analyzed (Participants) | 11 | 2 | 6 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 2 | 6 | 19
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.27 (9.00) | 32.50 (13.44) | 30.25 (10.66) | 30.48 (9.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 0 | 3 | 8
  Male | 6 | 2 | 3 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 9 | 2 | 6 | 17
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 2 | 6 | 19

OUTCOME MEASURES:

1. Primary Outcome: Reinforcing Effects (Pre-Alcohol Dose Consumption)
Description: The reinforcing effects of alcohol will be determined using a alcohol purchase task procedure in which subjects will report the number of alcohol drinks they would purchase across changes in price. The questions that were asked were completely hypothetical. The reinforcing effects are measured during experimental session maintenance on methylphenidate and placebo or duloxetine. These data represent "alpha", which a rate measure of sensitivity to changes in price: greater values represent great sensitivity to price changes. These data were collected prior to consumption of the alcohol dose. There is no minimum or maximum value.
Time Frame: Measured at each methylphenidate dose-level over approximately four weeks of participation.
Measure: Mean (95% Confidence Interval); unit: Units on a Theoretical Scale
Groups:
- Duloxetine 30 mg: Subjects received 30 mg of oral duloxetine one time daily. Alcohol: In each arm and during sessions, subjects will receive doses of alcohol designed to raise breath alcohol levels (BAL) to 0.03 g/dl.
  Duloxetine: Subjects will receive duloxetine capsules. Methylphenidate: Subjects will receive methylphenidate capsules.
Arm/Group | Placebo | Duloxetine 30 mg | Duloxetine (60 MG)
Number analyzed (Participants) | 9 | 2 | 6
Units on a Theoretical Scale
  Methylphenidate (0 mg) | 0.005 [0.0043 to 0.0057] | .01 [0.0078 to 0.012] | 0.007 [0.005 to 0.008]
  Methylphenidate (20 mg) | 0.005 [0.0041 to 0.0058] | .02 [0.014 to 0.020] | 0.007 [0.006 to 0.009]
  Methylphenidate (40 mg) | 0.005 [0.0041 to 0.0057] | 0.014 [0.012 to 0.018] | 0.007 [0.006 to 0.008]
  Methylphenidate (60 mg) | 0.005 [0.0041 to 0.0057] | .02 [0.012 to 0.020] | 0.008 [0.006 to 0.009]

2. Primary Outcome: Reinforcing Effects (Post-Alcohol Dose Consumption)
Description: The reinforcing effects of alcohol will be determined using a alcohol purchase procedure in which subjects will report the number of alcohol drinks they would purchase across changes in price. The questions that were asked were completely hypothetical. The reinforcing effects are measured during experimental session maintenance on methylphenidate and placebo or duloxetine. These data represent "alpha", which a rate measure of sensitivity to changes in price: greater values represent great sensitivity to price changes. These data were collected following consumption of the alcohol dose. There is no minimum or maximum value.
Time Frame: Measured at each methylphenidate dose-level over approximately four weeks of participation.
Measure: Mean (95% Confidence Interval); unit: Units on a Theoretical Scale
Arm/Group | Placebo | Duloxetine (30 MG) | Duloxetine (60 MG)
Number analyzed (Participants) | 9 | 2 | 6
Units on a Theoretical Scale
  Methylphenidate (0 mg) | 0.004 [0.0038 to 0.0052] | .01 [0.0075 to 0.010] | 0.006 [0.005 to 0.008]
  Methylphenidate (20 mg) | 0.005 [0.0041 to 0.0054] | .01 [0.010 to 0.013] | 0.007 [0.005 to 0.008]
  Methylphenidate (40 mg) | 0.005 [0.0039 to 0.0053] | .014 [0.011 to 0.017] | 0.006 [0.005 to 0.008]
  Methylphenidate (60 mg) | 0.005 [0.0044 to 0.0056] | .01 [0.010 to 0.016] | 0.009 [0.007 to 0.011]

3. Secondary Outcome: Visual Analog Scales of Alcohol Effects Following Methylphenidate (0 mg) Maintenance.
Description: Subjects will complete measures using visual analog scales rated from 0-100 mm to report alcohol effects during four experimental sessions. These items will ask about alcohol effects. Higher scores indicate greater effects. Data are presented as mean peak effect. Peak effect means the highest rated value (0 - 100 mm) following administration of oral alcohol
Time Frame: Measured at each methylphenidate dose-level over approximately four weeks of participation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Duloxetine (30 MG) | Duloxetine (60 MG)
Number analyzed (Participants) | 9 | 2 | 6
units on a scale
  Feel Drink | 15.89 (15.45) | 4.50 (2.12) | 22.00 (17.34)
  Feel High | 0.11 (0.33) | 1.00 (1.41) | 2.00 (3.95)
  Like Drink | 12.33 (16.08) | 4.50 (0.71) | 25.33 (20.30)
  Want Drink | 17.22 (17.48) | 7.50 (0.71) | 23.50 (20.42)

4. Secondary Outcome: Visual Analog Scales of Alcohol Effects Following Methylphenidate (20 mg) Maintenance.
Description: as for outcome 3
Time Frame: Measured at each methylphenidate dose-level over approximately four weeks of participation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Duloxetine (30 MG) | Duloxetine (60 MG)
Number analyzed (Participants) | 9 | 2 | 6
units on a scale
  Feel Drink | 17.44 (11.68) | 10.50 (6.36) | 28.50 (20.11)
  Feel High | 0.22 (0.67) | 1.50 (2.12) | 1.83 (4.02)
  Like Drink | 16.78 (23.55) | 9.50 (6.36) | 27.33 (22.14)
  Want Drink | 19.22 (19.57) | 15.50 (4.95) | 32.33 (24.66)

5. Secondary Outcome: Visual Analog Scales of Alcohol Effects Following Methylphenidate (40 mg) Maintenance.
Description: as for outcome 3
Time Frame: Measured at each methylphenidate dose-level over approximately four weeks of participation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Duloxetine (30 MG) | Duloxetine (60 MG)
Number analyzed (Participants) | 9 | 2 | 6
units on a scale
  Feel Drink | 10.67 (8.79) | 7.50 (2.12) | 20.17 (11.50)
  Feel High | 0.11 (0.33) | 1.00 (1.41) | 2.50 (4.18)
  Like Drink | 16.89 (21.97) | 10.00 (1.41) | 24.00 (18.28)
  Want Drink | 11.11 (12.58) | 15.00 (0.00) | 26.00 (27.31)

6. Secondary Outcome: Visual Analog Scales of Alcohol Effects Following Methylphenidate (60 mg) Maintenance.
Description: as for outcome 3
Time Frame: Measured at each methylphenidate dose-level over approximately four weeks of participation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Duloxetine (30 MG) | Duloxetine (60 MG)
Number analyzed (Participants) | 9 | 2 | 6
units on a scale
  Feel Drink | 12.67 (10.97) | 5.50 (2.12) | 17.17 (13.83)
  Feel High | 0.11 (0.33) | 1.00 (1.41) | 1.17 (2.40)
  Like Drink | 10.78 (12.77) | 8.00 (0.00) | 20.50 (21.14)
  Want Drink | 8.44 (13.60) | 15.00 (1.41) | 15.17 (11.48)

7. Secondary Outcome: Breath Alcohol Level
Description: Expired air samples for determining breath alcohol level (BAL) will be recorded during four experimental sessions. BALs were recorded as g/dl. Data are presented as mean peak effect. Peak effect means the highest rated value following administration of oral alcohol. Greater values of BAL represent more alcohol absorbed following consumption.
Time Frame: Measured at each methylphenidate dose-level over approximately four weeks of participation.
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | Placebo | Duloxetine (30 MG) | Duloxetine (60 MG)
Number analyzed (Participants) | 9 | 2 | 6
g/dl
  Methylphenidate (0 mg) | 0.026 (0.014) | 0.031 (0.006) | 0.029 (0.013)
  Methylphenidate (20 mg) | 0.024 (0.006) | 0.031 (0.004) | 0.042 (0.030)
  Methylphenidate (40 mg) | 0.024 (0.008) | 0.041 (0.006) | 0.034 (0.021)
  Methylphenidate (60 mg) | 0.026 (0.007) | 0.023 (0.005) | 0.037 (0.015)

8. Secondary Outcome: Systolic Blood Pressure
Description: Systolic blood pressure (millimeter of mercury) was recorded during four experimental sessions. Data are presented as mean peak effect. Peak effect means the highest rated value following administration of oral alcohol.
Time Frame: Measured at each methylphenidate dose-level over approximately four weeks of participation.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Placebo | Duloxetine (30 MG) | Duloxetine (60 MG)
Number analyzed (Participants) | 9 | 2 | 6
Millimeters of mercury
  Methylphenidate (0 mg) | 125.00 (13.65) | 129.00 (19.80) | 124.00 (8.90)
  Methylphenidate (20 mg) | 126.67 (12.35) | 140.00 (9.90) | 121.67 (6.53)
  Methylphenidate (40 mg) | 123.33 (10.39) | 130.00 (18.38) | 124.33 (8.73)
  Methylphenidate (60 mg) | 125.44 (12.17) | 131.50 (9.19) | 127.50 (11.98)

9. Secondary Outcome: Diastolic Blood Pressure
Description: Diastolic blood pressure (millimeter of mercury) was recorded during four experimental sessions. Data are presented as mean peak effect. Peak effect means the highest rated value following administration of oral alcohol.
Time Frame: Measured at each methylphenidate dose-level over approximately four weeks of participation.
Measure: Mean (Standard Deviation); unit: Millimeter of mercury
Arm/Group | Placebo | Duloxetine (30 MG) | Duloxetine (60 MG)
Number analyzed (Participants) | 9 | 2 | 6
Millimeter of mercury
  Methylphenidate (0 mg) | 73.56 (10.17) | 82.00 (12.73) | 77.67 (6.71)
  Methylphenidate (20 mg) | 74.00 (9.49) | 88.50 (6.36) | 77.00 (8.51)
  Methylphenidate (40 mg) | 74.22 (7.08) | 85.50 (9.19) | 80.33 (5.09)
  Methylphenidate (60 mg) | 74.00 (8.89) | 82.00 (8.49) | 80.50 (9.14)

10. Secondary Outcome: Heart Rate
Description: Heart rate (beats per minute) will be recorded during four experimental sessions. Data are presented as mean peak effect. Peak effect means the highest rated value following administration of oral alcohol.
Time Frame: Measured at each methylphenidate dose-level over approximately four weeks of participation.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | Duloxetine (30 MG) | Duloxetine (60 MG)
Number analyzed (Participants) | 9 | 2 | 6
Beats per minute
  Methylphenidate (0 mg) | 75.89 (11.47) | 66.50 (4.95) | 75.83 (11.41)
  Methylphenidate (20 mg) | 83.44 (12.63) | 80.50 (3.54) | 84.83 (11.43)
  Methylphenidate (40 mg) | 81.67 (7.48) | 73.50 (2.12) | 88.83 (13.01)
  Methylphenidate (60 mg) | 83.89 (13.04) | 80.50 (2.12) | 98.50 (21.72)

ADVERSE EVENTS:
Time Frame: Four weeks
Description: Please note that at the initial execution of the study, there were three duloxetine arms: 0, 30, and 60 mg/day. Two participants received 30 mg/day. However, to avoid the risk of HIPAA violation, data from these two participants will not be reported.
Groups:
- Duloxetine (60 MG): Subjects received 60 mg oral duloxetine one time daily.
  Alcohol: In each arm and during sessions, subjects will receive doses of alcohol designed to raise breath alcohol levels (BAL) to 0.03 g/dl.
  Duloxetine: Subjects will receive duloxetine capsules.
  Methylphenidate: Subjects will receive methylphenidate capsules.
Arm/Group | Placebo | Duloxetine (30 MG) | Duloxetine (60 MG)
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/2 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/2 | 0/6
Other Adverse Events (participants affected / at risk) | 11/11 | 2/2 | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=11) | Duloxetine (30 MG) (N=2) | Duloxetine (60 MG) (N=6)
Agitation (Nervous system disorders) | 3 (3) | 1 (1) | 1 (1)
Anxiety (Nervous system disorders) | 3 (3) | 2 (2) | 3 (3)
Body Aches (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 2 (2) | 2 (2)
Dry Mouth (General disorders) | 5 (5) | 1 (1) | 4 (4)
Ear Congestion (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0)
Change in Urination (General disorders) | 3 (3) | 0 (0) | 0 (0)
Headache (General disorders) | 4 (4) | 2 (2) | 3 (3)
Weakness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Loss of Voice (General disorders) | 0 (0) | 0 (0) | 2 (2)
Muscle Aches (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Nausea (General disorders) | 2 (2) | 2 (2) | 3 (3)
Nervousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Changes in Sexual Function (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Sleepiness/Dowsiness (General disorders) | 2 (2) | 2 (2) | 2 (2)
Sore Throat (General disorders) | 2 (2) | 2 (2) | 1 (1)
Stuffy/Runny nose (General disorders) | 2 (2) | 0 (0) | 0 (0)
Sweating (General disorders) | 1 (1) | 0 (0) | 3 (3)
Weight Change (General disorders) | 1 (1) | 0 (0) | 0 (0)
Unusual Bruising/Bleeding (General disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Restlessness (General disorders) | 3 (3) | 2 (2) | 3 (3)
Irritability (General disorders) | 3 (3) | 0 (0) | 0 (0)
Decreased Appetite (General disorders) | 4 (4) | 1 (1) | 2 (2)
Increased Appetite (General disorders) | 1 (1) | 1 (1) | 0 (0)
Insomnia (General disorders) | 2 (2) | 2 (2) | 4 (4)
Racing/Pounding Heart (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Itchness (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-31): https://cdn.clinicaltrials.gov/large-docs/03/NCT03575403/Prot_SAP_001.pdf
  • Informed Consent Form (2023-02-15): https://cdn.clinicaltrials.gov/large-docs/03/NCT03575403/ICF_002.pdf